CLINICAL TRIAL: NCT07264699
Title: Efficacy of Visually Guided Transversus Abdominis Plane (TAP) Block in Recovery After Laparoscopic Inguinal Hernia Repair (TAPP - Transabdominal Preperitoneal)
Brief Title: Visually Guided TAP Block in Laparoscopic TAPP Hernia Repair
Acronym: VIS-TAP-TAPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Responsible Party: Principal Investigator, Łukasz Dyśko, MD, University of Warmia and Mazury in Olsztyn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UWM-TAP-TAPP-2025; 19/2025/IX (Other: Ethics Committee Approval Number - Warmian-Masurian Chamber of Physicians in Olsztyn)
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Inguinal Hernia Repair; Postoperative Pain; TAP Block
Keywords: Inguinal hernia; TAPP; Laparoscopic hernia repair; TAP block; Transversus abdominis plane block; Multimodal analgesia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Dental Occlusion; Bupivacaine; tetra-4-amidinophenoxypropane

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel-group study comparing two interventions in patients undergoing elective laparoscopic inguinal hernia repair (TAPP). Participants will be randomly assigned in a 1:1 ratio to receive either a laparoscopically guided Transversus Abdominis Plane (TAP) block with 0.25% bupivacaine or no regional anesthesia. Both groups will receive identical perioperative care and standardized postoperative pain management. The design allows comparison of postoperative pain intensity and recovery outcomes between the TAP block and control groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study uses a single-blind design. Randomization is performed immediately before surgery using a concealed allocation sequence. The operating surgeons are aware of group assignment in order to perform the appropriate intervention (TAP block or none). Participants remain blinded to their allocation throughout the study period. Postoperative data, including pain intensity (VAS) and recovery parameters, are collected according to a standardized protocol by staff not involved in the randomization or intervention process to reduce potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block Group (Laparoscopic TAP Block with Bupivacaine) (Experimental): After pneumoperitoneum is established and the laparoscope is introduced, a bilateral Transversus Abdominis Plane (TAP) block is performed under direct laparoscopic vision. Using a needle and syringe, 20 ml of 0.25% bupivacaine is injected on each side, approximately 2 cm below the costal margin in the anterior axillary line. The correct placement of the local anesthetic is confirmed by the visible "Doyle's bulge sign." Patients receive standard general anesthesia and postoperative pain management identical to the control group.
  Interventions: Procedure: Laparoscopic Transversus Abdominis Plane (TAP) Block with Bupivacaine
- Control Group (No Regional Anesthesia - Standard Care) (No Intervention): Participants undergo standard laparoscopic inguinal hernia repair using the transabdominal preperitoneal (TAPP) technique without performing a TAP block or any other regional anesthesia. All patients receive the same standardized general anesthesia protocol and postoperative analgesic regimen as those in the experimental group.

INTERVENTIONS:
Procedure: Laparoscopic Transversus Abdominis Plane (TAP) Block with Bupivacaine — A bilateral Transversus Abdominis Plane (TAP) block is performed under direct laparoscopic vision after pneumoperitoneum is established. Using a needle and syringe, 20 ml of 0.25% bupivacaine is injected on each side, approximately 2 cm below the costal margin in the anterior axillary line. The correct spread of the local anesthetic is confirmed visually by observing the characteristic "Doyle's bulge sign." The procedure is performed before mesh placement during TAPP hernia repair. This technique allows direct visualization of the injection plane, increasing precision and safety compared with ultrasound-guided TAP blocks.
  Other Names: TAPP with TAP Block
  Arms: TAP Block Group (Laparoscopic TAP Block with Bupivacaine)

SUMMARY:
This prospective, randomized clinical study aims to evaluate the effectiveness of the Transversus Abdominis Plane (TAP) block performed under direct laparoscopic vision in reducing postoperative pain and improving recovery after laparoscopic inguinal hernia repair using the TAPP (Transabdominal Preperitoneal) technique.

The study will enroll 100 adult patients undergoing elective laparoscopic TAPP hernia repair at the University Clinical Hospital in Olsztyn, Poland. Participants will be randomly assigned to two equal groups. In the study group, a bilateral TAP block will be performed under direct vision using 20 ml of 0.25% bupivacaine on each side after establishing pneumoperitoneum. The control group will undergo the same surgical procedure without the TAP block.

All patients will receive standardized anesthesia and postoperative pain management according to hospital protocol. Postoperative pain intensity will be assessed using the Visual Analogue Scale (VAS) at 0, 6, and 12 hours after surgery. Additional data, such as time to mobilization, use of rescue analgesics, and occurrence of postoperative complications (hematoma, swelling, subcutaneous emphysema, transient muscle weakness), will also be recorded.

The primary goal of this study is to determine whether a laparoscopically guided TAP block can effectively reduce postoperative pain and improve recovery parameters following TAPP hernia repair. The results may help establish a simple, safe, and reproducible method of multimodal analgesia in minimally invasive inguinal hernia surgery.

DETAILED DESCRIPTION:
Inguinal hernia is one of the most common surgical conditions, affecting approximately 3% of the adult population. The only effective and lasting method of treatment is surgical repair. The laparoscopic transabdominal preperitoneal (TAPP) technique has become one of the most widely used minimally invasive approaches, offering reduced postoperative pain, shorter hospital stay, and faster return to daily activities compared with open repair. However, postoperative pain remains a relevant clinical problem and an important factor limiting early mobilization and recovery.

Multimodal analgesia is currently considered the standard approach for postoperative pain management. It combines systemic analgesics with regional anesthesia techniques. One of the increasingly used regional methods is the Transversus Abdominis Plane (TAP) block, which provides analgesia of the anterior abdominal wall by anesthetizing the intercostal, subcostal, iliohypogastric, and ilioinguinal nerves. The block can be performed under ultrasound guidance or, more recently, under direct laparoscopic vision, which improves safety and accuracy.

This single-center, prospective, randomized clinical study aims to assess the effect of a visually guided TAP block on postoperative pain and recovery after laparoscopic inguinal hernia repair (TAPP). The study will be conducted at the University Clinical Hospital in Olsztyn, Poland, between 2025 and 2027.

A total of 100 adult patients scheduled for elective laparoscopic TAPP hernia repair will be enrolled and randomly assigned (1:1) to one of two groups:

1. TAP Block Group (n = 50): After pneumoperitoneum is established and the laparoscope is introduced, a bilateral TAP block will be performed under direct vision. Using a needle and syringe, 20 ml of 0.25% bupivacaine (50 mg) will be injected approximately 2 cm below the costal margin in the anterior axillary line on both sides. Proper distribution of the local anesthetic will be confirmed visually by observing the characteristic elevation of the transversus abdominis muscle layer (known as the "Doyle's bulge sign").
2. Control Group (n = 50): The standard TAPP repair will be performed without additional regional anesthesia.

All patients will receive standardized general anesthesia and postoperative pain management. Analgesics will be administered according to a fixed schedule: metamizole 1.0 g orally at 6 and 12 hours after surgery. If needed, additional rescue medication will be provided: paracetamol 1.0 g orally for moderate pain (VAS < 6) or oxycodone 10 mg subcutaneously for severe pain (VAS > 6).

Pain intensity will be assessed using the Visual Analogue Scale (VAS) at 0, 6, and 12 hours after surgery, with separate evaluation for each surgical site (umbilical port, working trocar on the operated side, working trocar on the opposite side, operated groin, and operated testicle). Additional parameters include time to first mobilization, total analgesic consumption, and early postoperative recovery assessed with the Post Anesthesia Discharge Scoring System (PADSS). The occurrence of adverse events such as subcutaneous emphysema, hematoma, swelling, or transient lower limb weakness will also be recorded.

Patients with chronic pain syndromes, psychiatric disorders, alcohol or opioid dependence, recurrent hernias, or emergency indications will be excluded from the study. All participants will provide written informed consent before enrollment.

The collected data will be statistically analyzed to compare pain intensity, analgesic requirements, and recovery parameters between groups. The primary endpoint is postoperative pain intensity at 6 hours (VAS). Secondary endpoints include pain at 0 and 12 hours, time to mobilization, use of rescue analgesics, and adverse event rates.

The hypothesis of the study is that a laparoscopically guided TAP block significantly reduces postoperative pain intensity and improves recovery after laparoscopic TAPP hernia repair. The results of this study may contribute to the optimization of multimodal analgesia protocols in minimally invasive inguinal hernia surgery by introducing a simple, reproducible, and safe intraoperative analgesic technique.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Elective laparoscopic inguinal hernia repair using the TAPP (Transabdominal Preperitoneal) technique
* ASA physical status I-III
* Ability to provide written informed consent
* No contraindications to regional anesthesia or local anesthetic administration

Exclusion Criteria:

* Recurrent or strangulated inguinal hernia
* Emergency surgery
* Chronic pain syndromes or preoperative opioid use
* Known allergy or hypersensitivity to local anesthetics (bupivacaine or similar)
* Severe hepatic or renal impairment
* Psychiatric disorders or inability to provide informed consent
* Conversion to open surgery during the procedure
* Technical difficulties preventing TAP block administration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity (VAS score) at 6 hours after laparoscopic TAPP hernia repair | 6 hours postoperatively
  Pain intensity will be assessed using the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (worst pain imaginable). The measurement will focus on the operated area 6 hours after the completion of laparoscopic TAPP hernia repair. Pain will be recorded by trained nursing staff according to a standardized protocol. Scores from both groups (TAP block vs. control) will be compared to evaluate the analgesic effectiveness of the visually guided TAP block.

SECONDARY OUTCOMES:
Postoperative pain intensity (VAS score) at 0 and 12 hours after surgery | 0 and 12 hours after surgery
  Pain will be evaluated using the VAS scale (0-10) at 0 (immediately after surgery) and 12 hours postoperatively.
Time to first mobilization | Within 24 hours postoperatively
  The time (in hours) from the end of surgery to the patient's first ambulation will be recorded.
Need for rescue analgesia | First 12 hours after surgery
  Number of patients requiring additional analgesics (paracetamol or oxycodone) and total doses administered will be documented.
Postoperative recovery score (PADSS) | 6 hours after surgery
  Recovery will be assessed using the Post Anesthesia Discharge Scoring System (PADSS). A score ≥9 will indicate readiness for discharge.
Incidence of postoperative complications | Within 24 hours postoperatively
  Early postoperative complications such as hematoma, swelling, subcutaneous emphysema, or transient lower limb weakness will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marek Kowalczyk, PhD, MD, Principal Investigator — Clinic of Oncological and General Surgery, University Clinical Hospital in Olsztyn, Olsztyn, Poland
Locations (1):
- University Clinical Hospital in Olsztyn, Department of General and Oncological Surgery, Olsztyn, Warmisko-mazurskie, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center, investigator-initiated academic study involving a limited number of participants. The collected data include sensitive personal and clinical information that cannot be fully anonymized without compromising data integrity. Only aggregated, de-identified results will be published in peer-reviewed journals and conference presentations.